CLINICAL TRIAL: NCT02282527
Title: A Multi-center, Randomized, Double-blind, Crossover Study to Assess the Safety and Pharmacokinetics of Liquid Alpha₁-Proteinase Inhibitor (Human) Compared to Prolastin®-C in Subjects With Alpha₁-Antitrypsin Deficiency
Brief Title: A Study to Assess Safety and PK of Liquid Alpha₁-Proteinase Inhibitor (Human) in Treating Alpha₁-Antitrypsin Deficiency
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTI1402
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Alpha₁-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Sequence 1 (Other): Subjects were treated first with Liquid Alpha₁-PI and then treated with Prolastin-C
  Interventions: Biological: Liquid Alpha₁-PI; Biological: Prolastin-C
- Treatment Sequence 2 (Other): Subjects were treated first with Prolastin-C and then treated with Liquid Alpha₁-PI
  Interventions: Biological: Liquid Alpha₁-PI; Biological: Prolastin-C

INTERVENTIONS:
Biological: Liquid Alpha₁-PI — Liquid Alpha₁-PI, 60 mg/kg, 8 weekly intravenous infusions
Biological: Prolastin-C — Prolastin-C, 60 mg/kg, 8 weekly intravenous infusions

SUMMARY:
Grifols Therapeutics Inc. conducted a multi-center, randomized, double-blind, crossover study to evaluate the safety, immunogenicity, and pharmacokinetics (PK) of Liquid Alpha₁-PI compared to the currently licensed product, Prolastin-C, in subjects with Alpha₁-Antitrypsin Deficiency (AATD).

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 70 years of age, inclusive
* Had a diagnosis of congenital AATD
* Had a documented total alpha₁-PI level < 11 µM. If the total alpha₁-PI level had yet to be documented, a blood draw for total alpha₁-PI level was obtained at the Screening Visit
* Had a post-bronchodilator Forced expiratory volume in 1 second (FEV1) ≥ 30% and < 80% of predicted and FEV1/forced vital capacity (FVC) < 70%
* If the subject had received alpha₁-PI augmentation therapy of any kind, he/she must have been be willing to discontinue that treatment at the Week 1 (Baseline) Visit and remain off any kind of alpha₁-PI treatment, other than the investigational products for this study, while participating in the study

Exclusion Criteria:

* Subject had a moderate or severe pulmonary exacerbation during the 4 weeks before the Week 1 (Baseline) Visit
* History of lung or liver transplant
* Any lung surgery during the past 2 years (excluding lung biopsy)
* Liver cirrhosis confirmed by biopsy
* Elevated liver enzymes (aspartate transaminase [AST], alanine aminotransferase [ALT], and alkaline phosphatase [ALP]) equal to or greater than 2.5 times the upper limit of normal
* Severe concomitant disease (e.g., congestive heart failure, clinically significant pulmonary fibrosis, malignant disease [with the exception of skin cancers other than melanoma], history of acute hypersensitivity pneumonitis reaction, or current chronic hypersensitivity pneumonitis)
* Females who were pregnant, breastfeeding or, if of child-bearing potential, unwilling to practice a highly effective method of contraception (oral, injectable or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or abstinence) throughout the study
* Known previous infection with or clinical signs and symptoms consistent with current hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection
* Smoking during the past 6 months or a positive urine cotinine test at the Screening Visit that is due to smoking
* Participation in another investigational drug study within one month prior to the Week 1 (Baseline) Visit
* History of anaphylaxis or severe systemic response to any plasma-derived alpha1-PI preparation or other blood product(s)
* Use of systemic steroids above a stable dose equivalent to 5 mg/day prednisone (i.e.,10 mg every 2 days) within the 4 weeks prior to the Week 1 (Baseline) Visit inhaled steroids are not considered systemic steroids)
* Use of systemic or aerosolized antibiotics for an exacerbation within the 4 weeks prior to the Week 1 (Baseline) Visit
* Known selective or severe Immunoglobulin A (IgA) deficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - National Jewish Health, Denver, Colorado
  - University of Florida Gainesville, Gainesville, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Texas Health Science Center, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at 6 investigative centers in the US.
Groups:
- Liquid Alpha₁-PI/Prolastin-C: Subjects were treated first with Liquid Alpha₁-PI and then treated with Prolastin-C
  Liquid Alpha₁-PI: Liquid Alpha₁-PI, 60 mg/kg, 8 weekly intravenous infusions
  Prolastin-C: Prolastin-C, 60 mg/kg, 8 weekly intravenous infusions
- Prolastin-C/Liquid Alpha₁-PI: Subjects were treated first with Prolastin-C and then treated with Liquid Alpha₁-PI
  Prolastin-C: Prolastin-C, 60 mg/kg, 8 weekly intravenous infusions
  Liquid Alpha₁-PI: Liquid Alpha₁-PI, 60 mg/kg, 8 weekly intravenous infusions
Period: Overall Study
Arm/Group | Liquid Alpha₁-PI/Prolastin-C | Prolastin-C/Liquid Alpha₁-PI
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of home health aid | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liquid Alpha₁-PI/Prolastin-C | Prolastin-C/Liquid Alpha₁-PI | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (7.94) | 63.1 (5.93) | 61.9 (7.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Alpha1-PI concentration [Mean (Standard Deviation); unit: mg/mL] — Population: One subject in the Liquid Alpha₁-PI/Prolastin -C non-naïve population was missing baseline alpha₁-PI concentration due to sample instability.
  mg/mL
    Naive: number analyzed (Participants) | 1 | 3 | 4
    Naive | 0.31 (NA) — The standard deviation was not calculated as only 1 subject was assessed. | 0.21 (0.040) | 0.24 (0.059)
    Non-naive: number analyzed (Participants) | 14 | 13 | 27
    Non-naive | 0.72 (0.283) | 0.69 (0.215) | 0.70 (0.248)

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-7 Days) Based on Antigenic Content
Description: The primary PK objective of this study was to demonstrate the bioequivalence of Liquid Alpha₁-PI 60 mg/kg to Prolastin-C 60 mg/kg, as measured by AUC from 0 to 7 days (AUC0-7days) using an antigenic content assay of alpha₁-PI, at approximate steady state in subjects with AATD.
Time Frame: pre-dose, 0, 15 min, 30 min, 1 hour, 2 hours, 4 hours, 8 hours, 1 day, 2 days, 5 days, 7 days post dose
Measure: Mean (Standard Deviation); unit: mg*h/mL
Groups:
- Liquid Alpha₁-PI: Subjects treated with Liquid Alpha₁-PI in each treatment sequence
  Liquid Alpha₁-PI: Liquid Alpha1-PI, 60 mg/kg, 8 weekly intravenous infusions
- Prolastin-C: Subjects treated with Prolastin-C in each treatment sequence
  Prolastin-C: Prolastin-C, 60 mg/kg, 8 weekly intravenous infusions
Arm/Group | Liquid Alpha₁-PI | Prolastin-C
Number analyzed (Participants) | 30 | 28
mg*h/mL | 203.20 (23.041) | 198.38 (25.230)

2. Secondary Outcome: AUC(0-7 Days) Based on Functional Activity
Description: The exploratory PK objective of this study was to demonstrate the bioequivalence of Liquid Alpha₁-PI 60 mg/kg to Prolastin-C 60 mg/kg, as measured by AUC from 0 to 7 days (AUC 0-7 days) using a functional activity assay of alpha₁-PI, at approximate steady state in subjects with AATD.
Time Frame: pre-dose, 0, 15 min, 30 min, 1 hour, 2 hours, 4 hours, 8 hours, 1 day, 2 days, 5 days, 7 days post dose
Measure: Mean (Standard Deviation); unit: mg*h/mL
Groups:
- Liquid Alpha₁-PI: Subjects treated with Liquid Alpha₁-PI in each treatment sequence
  Liquid Alpha₁-PI: Liquid Alpha₁-PI, 60 mg/kg, 8 weekly intravenous infusions
Arm/Group | Liquid Alpha₁-PI | Prolastin-C
Number analyzed (Participants) | 30 | 28
mg*h/mL | 171.16 (28.764) | 168.50 (27.473)

3. Secondary Outcome: Number of Subjects With Immunogenicity Response
Description: Blood samples for immunogenicity testing were collected at Weeks 1 (Baseline), 9, 17, and 20. Any samples that tested positive for alpha₁-PI antibodies were tested for neutralizing antibodies and antibody titer. Immunogenicity testing was performed using validated assays in a multitiered approach. Samples collected at Week 1 (Baseline) and at Weeks 9 and 20 were tested for immunogenicity while samples collected at Week 17 were to be tested for immunogenicity only if deemed appropriate (eg, unexpected PK profile).
Time Frame: Weeks 1, 9, 17, and 20
Measure: Count of Participants; unit: Participants
Groups:
- Liquid Alpha₁-PI/Prolastin-C: Subjects were treated first with Liquid Alpha₁-PI and then treated with Prolastin-C
  Liquid Alpha₁-PI: Liquid Alpha1-PI, 60 mg/kg, 8 weekly intravenous infusions
  Prolastin-C: Prolastin-C, 60 mg/kg, 8 weekly intravenous infusions
Arm/Group | Liquid Alpha₁-PI/Prolastin-C | Prolastin-C/Liquid Alpha₁-PI
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Liquid Alpha₁-PI | Prolastin-C
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/31
Other Adverse Events (participants affected / at risk) | 9/32 | 3/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liquid Alpha₁-PI (N=32) | Prolastin-C (N=31)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liquid Alpha₁-PI (N=32) | Prolastin-C (N=31)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site may publish results from the study, after providing Sponsor at least 30 days notice prior to submitting a manuscript or other materials related to the study to any outside party. At Sponsor's request, Site will remove any any confidential information (other than study results), and incorporate all reasonable comments by Sponsor, or delay publication or presentation for a period of up to 120 days to allow Sponsor to protect its interests in any Sponsor's Inventions.